CLINICAL TRIAL: NCT00973700
Title: A Randomized, Open Label, Single Center, Dose- and Regimen-Ranging Study to Evaluate Immunogenicity, Safety and Tolerability of Different Formulations of an Adjuvanted and Non-Adjuvanted Egg-Derived, Inactivated Novel Swine Origin A/H1N1 Monovalent Subunit Influenza Virus Vaccine in Healthy Children and Adults Ages 3 to 64 Years
Brief Title: Safety and Immunogenicity of A/H1N1-SOIV (Swine Flu) Vaccine With and Without Adjuvant in Children, Adolescents and Adults (3 to 64 Years)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V112_04
Record Dates: First submitted 2009-09-02; First posted 2009-09-09 (Estimated); Results first posted 2011-05-23 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-10

CONDITIONS: Novel 2009 Influenza H1N1
Keywords: Swine Flu; Flu; Vaccine; Adjuvant
MeSH Terms: conditions — Orthomyxoviridae Infections; Influenza, Human

ARMS (5):
- 2x7.5adj (Experimental): Two doses of MF59 adjuvanted (adj) A/H1N1
  Interventions: Biological: MF59-eH1N1_f
- 7.5adj_1_8 (Experimental): MF59 adjuvanted (adj) A/H1N1 on days 1 and 8
  Interventions: Biological: MF59-eH1N1_f
- 7.5adj_1_22 (Experimental): MF59 adjuvanted (adj) A/H1N1 on study days 1 and 22
  Interventions: Biological: MF59-eH1N1_f
- 15_1_22 (Experimental): A/H1N1 on study days 1 and 22
  Interventions: Biological: eH1N1_f
- 2x15_1_22 (Experimental): Two doses of A/H1N1 (one in each arm) on study days 1 and 22
  Interventions: Biological: eH1N1_f

INTERVENTIONS:
Biological: MF59-eH1N1_f — MF59 adjuvanted (adj) egg-derived A/H1N1 with traces of Thiomersal
  Arms: 2x7.5adj; 7.5adj_1_22; 7.5adj_1_8
Biological: eH1N1_f — Unadjuvanted egg-derived A/H1N1 with traces of Thiomersal
  Arms: 15_1_22; 2x15_1_22

SUMMARY:
This study will evaluate the safety and immunogenicity of different combinations of A/H1N1 S-OIV (swine flu) vaccine in healthy young children, adolescents, and adults.

ELIGIBILITY:
Inclusion Criteria:

* Children, adolescents, and adults 3 to 64 years of age in good health as determined by medical history, physical assessment and clinical judgement of the investigator and without influenza within the past 6 months.

Exclusion Criteria:

* History of serious disease.
* History of serious reaction following administration of vaccine or hypersensitivity to vaccine components.
* Known or suspected impairment/alteration of immune function.
* Receipt or planned receipt of seasonal trivalent influenza vaccine within 1 week before or after each study vaccination.

For additional entry criteria, please refer to protocol.

Ages: 3 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 784 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Director — Novartis Vaccines
Locations (1):
- Instituto de Atencion Pediatrica, Avenida 0-2 Calle 22, Paseo Colon del Restaurante La, Bastilla 50 metros Sur, Edificio 5., San José, Costa Rica

REFERENCES:
- [Result] Arguedas A, Soley C, Abdelnour A, Sales V, Lindert K, Della Cioppa G, Clemens R; Costa Rican H1N1 Vaccine Study Group. Assessment of the safety, tolerability and kinetics of the immune response to A/H1N1v vaccine formulations with and without adjuvant in healthy pediatric subjects from 3 through 17 years of age. Hum Vaccin. 2011 Jan 1;7(1):58-66. doi: 10.4161/hv.7.1.13411. Epub 2011 Jan 1. PMID 21285531

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at one center in Costa Rica.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- 2x7.5adj: A/H1N1 7.5 mcg with MF59; two doses on day 1
- 7.5adj_1_8: A/H1N1 7.5 mcg with MF59; one dose on days 1 and 8
- 7.5adj_1_22: A/H1N1 7.5 mcg with MF59; one dose on days 1 and 22
- 15_1_22: A/H1N1 15 mcg no MF59; one dose on days 1 and 22
- 2x15_1_22: A/H1N1 15 mcg no MF59; two doses on days 1 and 22
Period: Overall Study
Arm/Group | 2x7.5adj | 7.5adj_1_8 | 7.5adj_1_22 | 15_1_22 | 2x15_1_22
Started | 56 | 56 | 168 | 336 | 168
Completed | 49 | 54 | 158 | 318 | 158
Not Completed | 7 | 2 | 10 | 18 | 10
Not completed — Withdrawal by Subject | 2 | 2 | 8 | 4 | 4
Not completed — Lost to Follow-up | 5 | 0 | 1 | 8 | 5
Not completed — Inappropriate enrolment | 0 | 0 | 0 | 4 | 0
Not completed — Unable to Classify | 0 | 0 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2x7.5adj | 7.5adj_1_8 | 7.5adj_1_22 | 15_1_22 | 2x15_1_22 | Total
Number analyzed (Participants) | 56 | 56 | 168 | 336 | 168 | 784
Age, Customized [Number; unit: subjects] — The number of participants analyzed for each outcome measure below is not the same with the numbers provided in the participant flow module as this number is based on the age and/or the group analyses.
  subjects
    3 to < 9 years | 0 (0) | 0 (0) | 56 (1.7) | 84 (1.7) | 56 (1.9) | 196
    9 to 17 years | 0 (0) | 0 (0) | 56 (2.5) | 84 (2.3) | 56 (2.5) | 196
    18 to 64 years | 56 (10.8) | 56 (11.1) | 56 (11.2) | 168 (11.7) | 56 (11.0) | 392
Sex/Gender, Customized [Number; unit: Subjects]
  Female (3 to <9 years) | 0 | 0 | 29 | 46 | 23 | 98
  Male (3 to < 9 years) | 0 | 0 | 27 | 38 | 33 | 98
  Female (9 to 17 years) | 0 | 0 | 40 | 40 | 30 | 110
  Male (9 to 17 years) | 0 | 0 | 16 | 44 | 26 | 86
  Female (18 to 64 years) | 33 | 40 | 29 | 96 | 29 | 227
  Male (18 to 64 years) | 23 | 16 | 27 | 72 | 27 | 165

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Seroconversion and HI Titer ≥1:40 in Children 3 to 17 Years of Age
Description: Seroconversion: The percentage of subjects with either a pre-vaccination HI titer < 1:10 and a post-vaccination HI titer >1:40 or a prevaccination HI titer >1:10 and a minimum four-fold rise in post-vaccination HI antibody titer.
  The analyses were performed on the Per-Protocol Set (PPS).
Time Frame: Day 1 to day 387
Population: The analysis was done on the per-protocol set.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 15_1_22
Number analyzed (Participants) | 149
Percentages of Subjects
  HI Titer ≥40 on day 1 | 26 [19 to 33]
  HI Titer ≥40 on day 22 | 83 [76 to 89]
  HI Titer ≥40 on day 29 | 95 [91 to 98]
  HI Titer ≥40 on day 43 | 92 [86 to 96]
  HI Titer ≥40 on day 217 (N=129) | 88 [81 to 93]
  HI Titer ≥40 on day 387 (N=136) | 80 [72 to 86]
  Seroconversion on day 22 | 79 [71 to 85]
  Seroconversion on day 29 | 92 [86 to 96]
  Seroconversion on day 43 | 87 [81 to 92]
  Seroconversion on day 217 (N=129) | 71 [62 to 78]
  Seroconversion on day 387 (N=136) | 63 [54 to 71]

2. Primary Outcome: Percentage of Subjects With Seroconversion and HI Titer ≥ 1:40 in Adults 18 to 64 Years of Age
Description: Seroconversion: The percentage of subjects with either a pre-vaccination HI titer < 1:10 and a post-vaccination HI titer >1:40 or a prevaccination HI titer >1:10 and a minimum four-fold rise in post-vaccination HI antibody titer.
  Analyses were performed on the Per-Protocol set (PPS).
Time Frame: Day 1 to day 387
Population: The analysis was done on the per-protocol set.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 15_1_22
Number analyzed (Participants) | 132
Percentages of Subjects
  HI Titer ≥40 on day 1 | 18 [12 to 26]
  HI Titer ≥40 on day 8 | 93 [87 to 97]
  HI Titer ≥40 on day 15 | 99 [96 to 100]
  HI Titer ≥40 on day 22 | 98 [95 to 100]
  HI Titer ≥40 on day 29 | 99 [96 to 100]
  HI Titer ≥40 on Day 43 | 100 [97 to 100]
  HI Titer ≥40 on Day 217 (N=111) | 91 [84 to 96]
  HI Titer ≥40 on Day 387 (N=120) | 84 [76 to 90]
  Seroconversion on day 8 | 86 [78 to 91]
  Seroconversion on day 15 | 94 [88 to 97]
  Seroconversion on day 22 | 94 [88 to 97]
  Seroconversion on day 29 | 95 [90 to 98]
  Seroconversion on day 43 | 95 [90 to 98]
  Seroconversion on day 217 (N=111) | 81 [73 to 88]
  Seroconversion on day 387 (N=120) | 75 [66 to 82]

3. Secondary Outcome: Age Distribution at Baseline
Time Frame: Baseline
Population: The overall number of baseline participants.
Measure: Mean (Standard Deviation); unit: years
Groups:
- 7.5adj_1_8; 7.5adj_1_22; 15_1_22; 2x15_1_22: A/H1N1 7.5 mcg with MF59; two doses on day 1
Arm/Group | 2x7.5adj | 7.5adj_1_8 | 7.5adj_1_22 | 15_1_22 | 2x15_1_22
Number analyzed (Participants) | 56 | 56 | 168 | 336 | 168
years
  3 to <9 years (N=0, 0, 56, 84, 56) | NA (NA) — Not Applicable (NA) as 0 subjects were in this category. | NA (NA) — Not Applicable (NA) as 0 subjects were in this category. | 5.5 (1.7) | 5.7 (1.7) | 5.4 (1.9)
  9 to 17 years (N=0, 0, 56, 84, 56) | NA (NA) — Not Applicable (NA) as 0 subjects were in this category. | NA (NA) — Not Applicable (NA) as 0 subjects were in this category. | 13.1 (2.5) | 12.8 (2.3) | 13.1 (2.5)
  18 to 64 years (N= 56, 56, 56, 168, 56) | 35.1 (10.8) | 38.6 (11.1) | 37.3 (11.2) | 37.0 (11.7) | 37.4 (11.0)

4. Secondary Outcome: Percentage of Subjects With Seroconversion and HI Titer ≥1:40, in 3 to <9 Years and 9 to 17 Years
Description: as for outcome 1
Time Frame: Day 1 to day 387
Population: The analysis is done on the per-protocol set.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 7.5adj_1_22 | 15_1_22 | 2x15_1_22
Number analyzed (Participants) | 91 | 149 | 99
Percentages of Subjects
  HI Titer ≥40 on day 1 (3 to <9 yrs; N=46,75,47) | 24 [13 to 39] | 23 [14 to 34] | 23 [12 to 38]
  HI Titer ≥40 on day 22 (3 to <9 yrs; N=46,75,47) | 93 [82 to 99] | 71 [59 to 81] | 79 [64 to 89]
  HI Titer ≥40 on day 29 (3 to < 9 yrs; N=46,75,47) | 100 [92 to 100] | 92 [83 to 97] | 96 [85 to 99]
  HI Titer ≥40 on day 43 (3 to < 9 yrs; N=46,75,47) | 100 [92 to 100] | 85 [75 to 92] | 96 [85 to 99]
  HI Titer ≥40 on day 217 (3 to < 9 yrs; N=41,66,40) | 100 [91 to 100] | 80 [69 to 89] | 78 [62 to 89]
  HI Titer ≥40 on day 387 (3 to < 9 yrs; N=43,70,42) | 93 [81 to 99] | 73 [61 to 83] | 62 [46 to 76]
  Seroconversion on day 22 (3 to <9 yrs; N=46,75,47) | 91 [79 to 98] | 69 [58 to 79] | 79 [64 to 89]
  Seroconversion on day 29 (3 to <9 yrs; N=46,75,47) | 98 [88 to 100] | 92 [83 to 97] | 96 [85 to 99]
  Seroconversion on day 43 (3 to <9 yrs; N=46,75,47) | 96 [85 to 99] | 84 [74 to 91] | 94 [82 to 99]
  Seroconversion on day 217 (3 to <9 yrs;N=41,66,40) | 88 [74 to 96] | 65 [52 to 76] | 65 [48 to 79]
  Seroconversion on day 387 (3 to <9 yrs;N=43,70,42) | 77 [61 to 88] | 56 [43 to 68] | 50 [34 to 66]
  HI Titer ≥40 on day 1 (9 to 17 yrs;N=45,74,52) | 42 [28 to 58] | 28 [19 to 40] | 33 [20 to 47]
  HI Titer ≥40 on day 22 (9 to 17 yrs; N=45,74,52) | 98 [88 to 100] | 96 [89 to 99] | 100 [93 to 100]
  HI Titer ≥40 on day 29 (9 to 17 yrs; N=45,74,52) | 100 [92 to 100] | 99 [93 to 100] | 100 [93 to 100]
  HI Titer ≥40 on day 43 (9 to 17 yrs; N=45,74,52) | 100 [92 to 100] | 99 [93 to 100] | 100 [93 to 100]
  HI Titer ≥40 on day 217 (9 to 17 yrs; N=37,63,45) | 100 [91 to 100] | 95 [87 to 99] | 98 [88 to 100]
  HI Titer ≥40 on day 387 (9 to 17 yrs; N=37,66,47) | 89 [75 to 97] | 88 [78 to 95] | 89 [77 to 96]
  Seroconversion on day 22 (9 to 17 yrs; N=45,74,52) | 87 [73 to 95] | 88 [78 to 94] | 94 [84 to 99]
  Seroconversion on day 29 (9 to 17 yrs; N=45,74,52) | 89 [76 to 96] | 92 [83 to 97] | 94 [84 to 99]
  Seroconversion on day 43 (9 to 17 yrs; N=45,74,52) | 84 [71 to 94] | 91 [81 to 96] | 92 [81 to 98]
  Seroconversion on day 217 (9 to 17 yrs;N=37,63,45) | 68 [50 to 82] | 76 [64 to 86] | 76 [60 to 87]
  Seroconversion on day 387 (9 to 17 yrs;N=37,66,47) | 59 [42 to 75] | 70 [57 to 80] | 70 [55 to 83]

5. Secondary Outcome: HI GMRs, in 3 to <9 Years and 9 to 17 Years
Description: Geometric Mean Ratios (GMRs) of hemagglutination inhibition (HI) antibody assay (ratio of post-vaccination versus pre-vaccination HI titers).
  The analyses were performed on the the per-protocol set (PPS).
Time Frame: Day 1 to day 387
Population: The analysis is done on the per-protocol set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | 7.5adj_1_22 | 15_1_22 | 2x15_1_22
Number analyzed (Participants) | 91 | 149 | 99
Ratio
  GMR on day 22 (3 to < 9 yrs; N=46,75,47) | 31 [19 to 50] | 12 [8.51 to 18] | 16 [10 to 26]
  GMR on day 29 (3 to < 9 yrs; N=46,75,47) | 169 [110 to 260] | 35 [24 to 49] | 53 [35 to 82]
  GMR on day 43 (3 to < 9 yrs; N=46,75,47) | 120 [75 to 192] | 22 [15 to 32] | 44 [27 to 69]
  GMR on day 217 (3 to <9 yrs; N=41,66,40) | 19 [12 to 30] | 7.79 [5.46 to 11] | 8.07 [5.11 to 13]
  GMR on day 387 (3 to <9 yrs; N=43,70,42) | 14 [8.27 to 24] | 6.9 [4.58 to 10] | 5.94 [3.5 to 10]
  GMR on day 22 (9 to 17 yrs; N=45,74,52) | 42 [24 to 74] | 52 [34 to 81] | 66 [39 to 111]
  GMR on day 29 (9 to 17 yrs; N=45,74,52) | 63 [36 to 109] | 70 [45 to 108] | 79 [47 to 132]
  GMR on day 43 (9 to 17 yrs; N=45,74,52) | 44 [25 to 77] | 48 [31 to 75] | 59 [35 to 100]
  GMR on day 217 (9 to 17 yrs; N=37,63,45) | 10 [5.66 to 18] | 17 [11 to 26] | 13 [7.92 to 23]
  GMR on day 387 (9 to 17 yrs; N=37,66,47) | 7.22 [3.77 to 14] | 16 [9.53 to 25] | 13 [7.53 to 24]

6. Secondary Outcome: HI GMR, in Adults 18 to 64 Years
Description: Geometric Mean Ratios (GMRs) of hemagglutination inhibition (HI) antibody assay (ratio of post-vaccination versus pre-vaccination HI titers).
  The analyses were performed on the Per-Protocol Set (PPS).
Time Frame: Day 1 to day 387
Population: The analysis is done on the per-protocol set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | 2x7.5adj | 7.5adj_1_8 | 7.5adj_1_22 | 15_1_22 | 2x15_1_22
Number analyzed (Participants) | 41 | 45 | 45 | 132 | 47
Ratio
  GMR on day 8 | 48 [28 to 85] | 35 [21 to 60] | 57 [33 to 97] | 43 [32 to 59] | 63 [37 to 106]
  GMR on day 15 | 115 [70 to 189] | 181 [113 to 292] | 200 [124 to 322] | 138 [104 to 182] | 123 [77 to 197]
  GMR on day 22 | 79 [48 to 130] | 100 [63 to 160] | 123 [77 to 197] | 85 [64 to 111] | 72 [45 to 113]
  GMR on day 29 | 56 [35 to 89] | 76 [49 to 118] | 160 [103 to 248] | 83 [64 to 107] | 66 [43 to 101]
  GMR on day 43 | 44 [27 to 71] | 64 [40 to 101] | 101 [63 to 161] | 76 [58 to 100] | 65 [41 to 102]
  GMR on day (N=0,0,35,111,34) | NA [NA to NA] — Zero subjects were enrolled in this group. | NA [NA to NA] — Zero subjects were enrolled in this group. | 30 [18 to 48] | 16 [12 to 20] | 16 [10 to 27]
  GMR on day 387 (N=38,40,38,120,42) | 6.61 [3.92 to 11] | 11 [6.81 to 19] | 21 [12 to 36] | 12 [8.99 to 16] | 9.21 [5.61 to 15]

7. Secondary Outcome: Percentage of Subjects With Seroconversion and HI Titer ≥1:40, in Adults 18 to 64 Years
Description: as for outcome 1
Time Frame: 7 days and 21 days after each vaccination
Population: The analysis is done on the per-protocol set.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 2x7.5adj | 7.5adj_1_8 | 7.5adj_1_22 | 15_1_22 | 2x15_1_22
Number analyzed (Participants) | 41 | 45 | 45 | 132 | 47
Percentages of Subjects
  HI Titer ≥40 on day 8 | 100 [91 to 100] | 91 [79 to 98] | 96 [85 to 99] | 93 [87 to 97] | 96 [85 to 99]
  HI Titer ≥40 on day 15 | 100 [91 to 100] | 100 [92 to 100] | 98 [88 to 100] | 99 [96 to 100] | 100 [92 to 100]
  HI Titer ≥40 on day 22 | 100 [91 to 100] | 98 [88 to 100] | 98 [88 to 100] | 98 [95 to 100] | 98 [89 to 100]
  HI Titer ≥40 on day 29 | 100 [91 to 100] | 98 [88 to 100] | 100 [92 to 100] | 99 [96 to 100] | 100 [92 to 100]
  HI Titer ≥40 on day 43 | 98 [87 to 100] | 100 [92 to 100] | 98 [88 to 100] | 100 [97 to 100] | 100 [92 to 100]
  HI Titer ≥40 on day 217 (N=0,0,35,111,34) | NA [NA to NA] — No subjects were analyzed for this group. | NA [NA to NA] — No subjects were analyzed for this group. | 97 [85 to 100] | 91 [84 to 96] | 97 [85 to 100]
  HI Titer ≥40 on day 387 (N=38,40,38,120,42) | 76 [60 to 89] | 90 [76 to 97] | 92 [79 to 98] | 84 [76 to 90] | 83 [69 to 93]
  Seroconversion on day 8 | 95 [83 to 99] | 80 [65 to 90] | 93 [82 to 99] | 86 [78 to 91] | 94 [82 to 99]
  Seroconversion on day 15 | 98 [87 to 100] | 100 [92 to 100] | 98 [88 to 100] | 94 [88 to 97] | 98 [89 to 100]
  Seroconversion on day 22 | 95 [83 to 99] | 91 [79 to 98] | 96 [85 to 99] | 94 [88 to 97] | 96 [85 to 99]
  Seroconversion on day 29 | 95 [83 to 99] | 93 [82 to 99] | 98 [88 to 100] | 95 [90 to 98] | 98 [89 to 100]
  Seroconversion on day 43 | 85 [71 to 94] | 93 [82 to 99] | 96 [85 to 99] | 95 [90 to 98] | 98 [89 to 100]
  Seroconversion on day 217 (N=0,0,35,111,34) | NA [NA to NA] — No subjects were analyzed for this group. | NA [NA to NA] — No subjects were analyzed for this group. | 94 [81 to 99] | 81 [73 to 88] | 88 [73 to 97]
  Seroconversion on day 387 (N=38,40,38,120,42) | 66 [49 to 80] | 80 [64 to 91] | 87 [72 to 96] | 75 [66 to 82] | 69 [53 to 82]
  HI Titer ≥40 on day 1 | 20 [9 to 35] | 22 [11 to 37] | 13 [5 to 27] | 18 [12 to 26] | 21 [11 to 36]

8. Secondary Outcome: Number of Subjects With at Least One Reactogenicity Sign, in 3 to <9 Years of Age
Description: Number of subjects with specified solicited local and systemic reactions in adult subjects (3 to <9 years of age).
  Postvac: postvaccination; Analges: analgesics; Antipyr: antipyretics. The analyses were performed on the safety set. Note: 1) postvac 1 = after the first vaccination and 2) postvac 2 = after the second vaccination
Time Frame: 7 days after each vaccination
Population: The analysis is done on the safety set.
Measure: Number; unit: Number of subjects
Arm/Group | 7.5adj_1_22 | 15_1_22 | 2x15_1_22
Number analyzed (Participants) | 55 | 84 | 54
Number of subjects
  Local Reactions postvac. 1 | 25 | 31 | 20
  Erythema postvac. 1 | 1 | 0 | 0
  Induration postvac. 1 | 0 | 3 | 1
  Swelling postvac. 1 | 3 | 4 | 3
  Tenderness postvac. 1 | 21 | 23 | 17
  Pain postvac. 1 | 21 | 25 | 17
  Systemic Reaction postvac. 1 | 24 | 28 | 17
  Headache postvac. 1 | 7 | 12 | 9
  Fatigue postvac. 1 | 6 | 8 | 5
  Myalgia postvac. 1 | 4 | 8 | 6
  Arthralgia postvac. 1 | 0 | 2 | 2
  Chills postvac. 1 | 3 | 1 | 2
  Nausea postvac. 1 | 5 | 7 | 4
  Vomiting postvac. 1 | 0 | 1 | 2
  Diarrhea postvac. 1 | 0 | 0 | 1
  Other Reactions postvac. 1 | 10 | 10 | 6
  Analges/Antipyr Used postvac. 1 (N=55, 83, 54) | 9 | 8 | 6
  Stayed Home postvac.1(N=55,83,54) | 1 | 2 | 0
  Body Temp > 40 C postvac.1 | 0 | 0 | 0
  Local Reactions postvac. 2 (N=55, 83, 54) | 20 | 29 | 21
  Erythema postvac. 2 (N=55, 83, 54) | 3 | 1 | 1
  Induration postvac. 2 (N=55, 83, 54) | 8 | 1 | 2
  Swelling postvac. 2 (N=55, 83, 54) | 8 | 0 | 2
  Tenderness postvac. 2 (N=55, 83, 54) | 15 | 27 | 16
  Pain postvac. 2 (N=55, 83, 54) | 18 | 23 | 19
  Systemic Reaction postvac. 2 (N=55, 83, 54) | 13 | 22 | 18
  Headache postvac. 2 (N=55, 83, 54) | 5 | 12 | 3
  Fatigue postvac. 2 (N=55, 83, 54) | 1 | 5 | 2
  Myalgia postvac. 2 (N=55, 83, 54) | 3 | 2 | 5
  Arthralgia postvac. 2 (N=55, 83, 54) | 0 | 2 | 5
  Chills postvac. 2 (N=55, 83, 54) | 2 | 2 | 1
  Nausea postvac. 2 (N=55, 83, 54) | 5 | 5 | 1
  Vomiting postvac. 2 (N=55, 83, 54) | 0 | 1 | 3
  Diarrhea postvac. 2 (N=55, 83, 54) | 0 | 1 | 2
  Other Reactions postvac. 2 (N=55, 82, 54) | 5 | 7 | 7
  Analges/Antipyr Used postvac. 2 (N=55, 83, 54) | 4 | 6 | 7
  Stayed Home postvac. 2 (N=55, 82, 54) | 1 | 2 | 0
  Body Temp > 40 C postvac. 2 (N=55, 83, 54) | 0 | 0 | 0

9. Secondary Outcome: Number of Subjects With at Least One Reactogenicity Sign, in 9 to 17 Years of Age
Description: Number of subjects with specified solicited local and systemic reactions in adult subjects (9 to 17 years of age).
  Postvac: postvaccination Analges: analgesics Antipyr: antipyretics The analyses were performed on the safety set.
  Note: 1) postvac 1 = after the first vaccination and 2) postvac 2 = after the second vaccination.
Time Frame: 7 days after each vaccination
Population: The analysis is done on the safety set.
Measure: Number; unit: Number of subjects
Arm/Group | 7.5adj_1_22 | 15_1_22 | 2x15_1_22
Number analyzed (Participants) | 53 | 84 | 57
Number of subjects
  Local Reactions postvac. 1 | 37 | 36 | 29
  Erythema postvac. 1 | 1 | 1 | 0
  Induration postvac. 1 | 1 | 6 | 1
  Swelling postvac. 1 | 1 | 4 | 3
  Tenderness postvac. 1 | 26 | 23 | 21
  Pain postvac. 1 | 32 | 30 | 25
  Systemic Reaction postvac. 1 | 24 | 36 | 16
  Headache postvac. 1 | 17 | 20 | 8
  Fatigue postvac. 1 | 9 | 13 | 11
  Myalgia postvac. 1 | 11 | 15 | 11
  Arthralgia postvac. 1 | 2 | 2 | 0
  Chills postvac. 1 | 1 | 2 | 1
  Nausea postvac. 1 | 3 | 7 | 5
  Vomiting postvac. 1 | 0 | 1 | 0
  Diarrhea postvac. 1 | 2 | 0 | 0
  Other Reactions postvac. 1 | 11 | 10 | 8
  Analgesic/Antipyretic Used postvac. 1 | 10 | 10 | 7
  Stayed Home postvac. 1 | 2 | 1 | 2
  Body Temp > 40 C postvac. 1 | 0 | 0 | 0
  Local Reactions postvac. 2 (N=52, 84, 55) | 31 | 36 | 27
  Erythema postvac. 2 (N=52, 84, 55) | 0 | 3 | 1
  Induration postvac. 2 (N=52, 84, 55) | 2 | 3 | 4
  Swelling postvac. 2 (N=52, 84, 55) | 2 | 5 | 3
  Tenderness postvac. 2 (N=52, 84, 55) | 20 | 25 | 25
  Pain postvac. 2 (N=52, 84, 55) | 27 | 30 | 26
  Systemic Reaction postvac. 2 (N=52, 84, 55) | 18 | 29 | 14
  Headache postvac. 2 (N=52, 84, 55) | 12 | 16 | 8
  Fatigue postvac. 2 (N=52, 84, 55) | 3 | 6 | 9
  Myalgia postvac. 2 (N=52, 84, 55) | 8 | 9 | 7
  Arthralgia postvac. 2 (N=52, 84, 55) | 0 | 4 | 4
  Chills postvac. 2 (N=52, 84, 55) | 2 | 2 | 3
  Nausea postvac. 2 (N=52, 84, 55) | 3 | 7 | 2
  Vomiting postvac. 2 (N=52, 84, 55) | 1 | 0 | 0
  Diarrhea postvac. 2 (N=52, 84, 55) | 2 | 3 | 0
  Other Reactions postvac. 2 (N=52, 84, 55) | 1 | 10 | 4
  Analges/Antipyr Used postvac. 2 (N=52, 84, 55) | 1 | 9 | 4
  Stayed Home postvac. 2 (N=52, 84, 55) | 0 | 1 | 0
  Body Temp > 40 C postvac. 2 (N=52, 84, 55) | 0 | 0 | 0

10. Secondary Outcome: Number of Subjects With at Least One Reactogenicity Sign, in 18 to 64 Years of Age
Description: Number of subjects with specified solicited local and systemic reactions in adult subjects (18 to 64 years of age).
  Note: 1) postvac. 1 = after the first vaccination and 2) postvac. 2 = after the second vaccination.
  The analyses were performed on the safety set.
Time Frame: 7 days after each vaccination
Population: The analysis is done on the safety set.
Measure: Number; unit: Number of subjects
Arm/Group | 2x7.5adj | 7.5adj_1_8 | 7.5adj_1_22 | 15_1_22 | 2x15_1_22
Number analyzed (Participants) | 54 | 56 | 56 | 159 | 54
Number of subjects
  Local Reactions postvac. 1 | 39 | 26 | 38 | 56 | 19
  Erythema postvac. 1 | 3 | 0 | 2 | 2 | 1
  Induration postvac. 1 | 5 | 4 | 5 | 6 | 3
  Swelling postvac. 1 | 3 | 3 | 5 | 4 | 2
  Tenderness postvac. 1 | 33 | 21 | 26 | 35 | 14
  Pain postvac. 1 | 36 | 23 | 32 | 41 | 16
  Systemic Reaction postvac. 1 | 34 | 31 | 31 | 71 | 22
  Headache postvac. 1 | 26 | 18 | 22 | 42 | 12
  Fatigue postvac. 1 | 17 | 16 | 16 | 32 | 15
  Myalgia postvac. 1 | 21 | 13 | 16 | 28 | 12
  Arthralgia postvac. 1 | 4 | 1 | 6 | 10 | 2
  Chills postvac. 1 | 4 | 3 | 6 | 6 | 4
  Nausea postvac. 1 | 7 | 9 | 8 | 16 | 13
  Vomiting postvac. 1 | 0 | 0 | 0 | 1 | 1
  Diarrhea postvac. 1 | 2 | 1 | 0 | 8 | 3
  Other Reactions postvac. 1 | 14 | 7 | 12 | 13 | 5
  Analgesic/Antipyretic Used postvac. 1 | 14 | 6 | 12 | 13 | 4
  Stayed Home postvac. 1 (N=53,55,56,157,54) | 2 | 1 | 2 | 0 | 1
  Body Temp > 40 C postvac. 1 | 0 | 0 | 0 | 0 | 0
  Local Reactions postvac. 2 (N=0,55,56,158,53) | 0 | 21 | 28 | 56 | 17
  Erythema postvac. 2 (N=0,55,56,158,53) | 0 | 1 | 2 | 5 | 1
  Induration postvac. 2 (N=0,55,56,158,53) | 0 | 3 | 4 | 4 | 3
  Swelling postvac. 2 (N=0,55,56,158,53) | 0 | 2 | 5 | 7 | 5
  Tenderness postvac. 2 (N=0,55,56,157853) | 0 | 16 | 24 | 48 | 16
  Pain postvac. 2 (N=0,55,56,158,53) | 0 | 19 | 24 | 45 | 15
  Systemic Reaction postvac. 2 (N=0,55,56,158,53) | 0 | 26 | 28 | 53 | 14
  Headache postvac. 2 (N=0,55,56,158, 53) | 0 | 18 | 18 | 25 | 11
  Fatigue postvac. 2 (N=0,55,56,158, 53) | 0 | 14 | 13 | 24 | 10
  Myalgia postvac. 2 (N=0,55,56,158, 53) | 0 | 9 | 14 | 26 | 7
  Arthralgia postvac. 2 (N=0,55,56,158, 53) | 0 | 5 | 7 | 16 | 4
  Chills postvac. 2 (N=0,55,56,158, 53) | 0 | 8 | 5 | 5 | 8
  Nausea postvac. 2 (N=0,55,56,158, 53) | 0 | 8 | 5 | 7 | 3
  Vomiting postvac. 2 (N=0,55,56,158, 53) | 0 | 1 | 0 | 2 | 1
  Diarrhea postvac. 2 (N=0,55,56,158, 53) | 0 | 1 | 0 | 4 | 1
  Other Reactions postvac. 2 (N=0,55,56,158, 53) | 0 | 8 | 7 | 11 | 7
  Analgesi/Antipyr Used postvac 2 (N=0,55,56,158,53) | 0 | 7 | 7 | 11 | 6
  Stayed Home postvaccination 2 (N=0,53,0,156,53) | 0 | 2 | 0 | 1 | 2
  Body Temp > 40 C postvac. 2 (N=0,55,56,158,53) | 0 | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) and serious adverse events were collected throughout the duration of the study (day 1 to day 387).
Description: Data provided in Other Adverse Events (>5%) were collected. The data included solicited local and systemic reactions that persisted for more than 7 days after each study vaccination. The number of participants at risk is not the same with the numbers provided in the participant flow module as these numbers are analyzed by age and group.
Groups:
- 2x7.5adj (18 to 64 Yrs): A/H1N1 7.5 mcg with MF59; two doses on day 1
- 7.5adj_1_8 (18 to 64 Yrs): A/H1N1 7.5 mcg with MF59; one dose on days 1 and 8
- 7.5adj_1_22 (18-64 Yrs); 7.5adj_1_22 (9 to 17 Yrs); 7.5adj_1_22 (3 to <9 Yrs): A/H1N1 7.5 mcg with MF59; one dose on days 1 and 22
- 15_1_22 (18 to 64 Yrs); 15_1_22 (9 to 17 Yrs); 15_1_22 (3 to <9 Yrs): A/H1N1 15 mcg no MF59; one dose on days 1 and 22
- 2x15_1_22 (18 to 64 Yrs); 2x15_1_22 (9 to 17 Yrs); 2x15_1_22 (3 to <9 Yrs): A/H1N1 15 mcg no MF59; two doses on days 1 and 22
Arm/Group | 2x7.5adj (18 to 64 Yrs) | 7.5adj_1_8 (18 to 64 Yrs) | 7.5adj_1_22 (18-64 Yrs) | 15_1_22 (18 to 64 Yrs) | 2x15_1_22 (18 to 64 Yrs) | 7.5adj_1_22 (9 to 17 Yrs) | 15_1_22 (9 to 17 Yrs) | 2x15_1_22 (9 to 17 Yrs) | 7.5adj_1_22 (3 to <9 Yrs) | 15_1_22 (3 to <9 Yrs) | 2x15_1_22 (3 to <9 Yrs)
Serious Adverse Events (participants affected / at risk) | 2/54 | 0/56 | 1/56 | 4/159 | 1/54 | 1/53 | 1/84 | 0/57 | 2/55 | 0/84 | 0/54
Other Adverse Events (participants affected / at risk) | 49/54 | 41/56 | 48/56 | 119/159 | 35/54 | 46/53 | 67/84 | 43/57 | 40/55 | 61/84 | 41/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2x7.5adj (18 to 64 Yrs) (N=54) | 7.5adj_1_8 (18 to 64 Yrs) (N=56) | 7.5adj_1_22 (18-64 Yrs) (N=56) | 15_1_22 (18 to 64 Yrs) (N=159) | 2x15_1_22 (18 to 64 Yrs) (N=54) | 7.5adj_1_22 (9 to 17 Yrs) (N=53) | 15_1_22 (9 to 17 Yrs) (N=84) | 2x15_1_22 (9 to 17 Yrs) (N=57) | 7.5adj_1_22 (3 to <9 Yrs) (N=55) | 15_1_22 (3 to <9 Yrs) (N=84) | 2x15_1_22 (3 to <9 Yrs) (N=54)
appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
rhinoplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — This AE was reported in the Adults (18 to 64 years of age) under group 2x15_1_22.
Precocious Puberty (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
sexual abuse (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
high risk pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hysterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2x7.5adj (18 to 64 Yrs) (N=54) | 7.5adj_1_8 (18 to 64 Yrs) (N=56) | 7.5adj_1_22 (18-64 Yrs) (N=56) | 15_1_22 (18 to 64 Yrs) (N=159) | 2x15_1_22 (18 to 64 Yrs) (N=54) | 7.5adj_1_22 (9 to 17 Yrs) (N=53) | 15_1_22 (9 to 17 Yrs) (N=84) | 2x15_1_22 (9 to 17 Yrs) (N=57) | 7.5adj_1_22 (3 to <9 Yrs) (N=55) | 15_1_22 (3 to <9 Yrs) (N=84) | 2x15_1_22 (3 to <9 Yrs) (N=54)
nasopharyngitis (Infections and infestations) | 10 (11) | 6 (7) | 8 (8) | 24 (26) | 6 (7) | 7 (7) | 12 (15) | 11 (12) | 4 (6) | 17 (20) | 11 (15)
upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 5 (6) | 6 (7) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 4 (5) | 7 (9) | 6 (7)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 8 (9) | 3 (3) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 6 (7) | 4 (5)
headache (Nervous system disorders) | 27 (31) | 21 (49) | 27 (57) | 56 (91) | 17 (30) | 21 (39) | 29 (48) | 11 (22) | 11 (12) | 21 (31) | 11 (15)
myalgia (Musculoskeletal and connective tissue disorders) | 21 (28) | 17 (25) | 21 (34) | 42 (73) | 17 (22) | 18 (22) | 20 (26) | 14 (22) | 5 (8) | 10 (12) | 9 (13)
injection site erythema (General disorders) | 3 (5) | 1 (1) | 3 (4) | 6 (7) | 2 (3) | 1 (1) | 4 (4) | 1 (1) | 3 (4) | 1 (1) | 1 (1)
injection site pain (General disorders) | 39 (130) | 31 (79) | 42 (113) | 79 (173) | 23 (108) | 42 (116) | 52 (117) | 37 (160) | 32 (75) | 43 (102) | 29 (116)
injection site swelling (General disorders) | 1 (2) | 2 (2) | 2 (2) | 5 (5) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 2 (2)
nausea (Gastrointestinal disorders) | 7 (7) | 13 (23) | 11 (17) | 21 (28) | 5 (8) | 6 (6) | 12 (16) | 6 (11) | 8 (10) | 10 (14) | 5 (5)
pyrexia (General disorders) | 2 (2) | 4 (5) | 6 (8) | 12 (13) | 2 (2) | 3 (4) | 3 (3) | 6 (8) | 8 (8) | 10 (13) | 10 (12)
fatigue (General disorders) | 17 (20) | 20 (34) | 21 (36) | 45 (73) | 18 (30) | 11 (13) | 15 (23) | 14 (26) | 6 (7) | 11 (16) | 6 (9)
arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6) | 10 (14) | 24 (32) | 4 (7) | 2 (2) | 5 (7) | 5 (5) | 0 (0) | 4 (4) | 7 (7)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 1 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 5 (5)
dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
chills (General disorders) | 4 (5) | 9 (11) | 8 (12) | 10 (12) | 11 (14) | 3 (3) | 4 (4) | 4 (5) | 4 (6) | 2 (3) | 2 (3)
diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (4) | 1 (1) | 13 (13) | 3 (5) | 4 (4) | 5 (5) | 0 (0) | 1 (1) | 3 (3) | 5 (5)
tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (3) | 6 (6)
varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
backpain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (4) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No